CLINICAL TRIAL: NCT06822140
Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation on Motor and Cognitive Deficits After Ischemic Stroke
Brief Title: Effect of Vagus Nerve Stimulation Via the Outer Ear on Motor and Cognitive Deficits After Ischemic Stroke
Acronym: EVAMOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rheinburg-Klinik (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-D0114
Record Dates: First submitted 2025-02-05; First posted 2025-02-12 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Ischemic Stroke; Motor Deficits; Cognitive Impairment; Vagus Nerve Stimulation
MeSH Terms: conditions — Ischemic Stroke; Neurologic Manifestations; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VNS group (Experimental)
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- control group (Sham Comparator)
  Interventions: Device: sham-stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — Stimulation parameters:
  * Stimulating side: ipsilateral to the infarcted brain hemisphere
  * Location of pStimulation: Cymba conchae
  * Impulse shape: bi-phasic
  * Impulse intensity: at least 0.5 mA (max. 2.0 mA).
  * Impulse duration: 28 sec on, 32 sec off
  * Impulse frequency: 20-30 Hz.
  Arms: VNS group
Device: sham-stimulation — An electrode is only attached to the ear without applying electrical impulses.
  Arms: control group

SUMMARY:
The goal of this clinical trial is to learn if transcutaneous auricular vagus nerve stimulation (taVNS) works to treat motor and neurocognitive deficits after ischemic stroke when applied within 30 days after onset of stroke.

The main questions it aims to answer are:

* Does tVNS improve motor deficits measured by the Fugl-Mayer assessment after ischemic stroke?
* Does tVNS ameliorate stroke-related cognitive impairment? Researchers will compare tVNS to a placebo (sham stimulation, i.e. an electrode is fixed on the ear without applying electrical impulses ) to see if tVNS works to treat motor and cognitive deficits after stroke .

Participants will:

* Receive tVNS or sham stimulation for 30 minutes 5 days a week during 5 weeks after ischemic stroke
* Receive smotor and cognitive training during the tVNS or sham stimulation
* Will take part on a standardized stroke rehabilitation program during the 5 weeks in a rehabilitation clinic.

DETAILED DESCRIPTION:
Study participants will undergo pre-evaluation and receive information within the first 7 days after admission to the Rheinburg-Klinik (Visit 0). During these 7 days, study participants will be randomly (1:1) allocated to the intervention group (taVNS) or control group (sham-stimulation) and will be clinically examined (Visit 1). At Visit 2 (≤7 days after admission), baseline assessments will be performed. During the intervention period, (week 2 to 6 after admission), either taVNS or sham-stimulation will be conducted for 30 minutes per day at 5 days per week for 5 weeks, paired with cognitive and motor training. Participants will be blinded to treatment. Standardized rehabilitation measures according to the clinic standards will be performed in both groups during the study period. All study participants will be monitored by recording an ECG during intervention/sham-stimulation. Before and after intervention/sham-stimulation an EEG will be conducted. After intervention, i.e., at the end of week 6, the same assessments as at baseline will be repeated (Visit 3). A follow up visit will take place 6 months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Onset of stroke ≥15 days and ≤30 days after randomization
* Ischemic stroke in the anterior cerebral circulation detected by MR imaging or computer tomography
* National Institutes of Health Stroke Scale (NIHSS) score ≥3 points
* Montreal Cognitive Assessment (MoCA) score ≤ 26 points
* First ever stroke
* Right-handed
* Ability to participate in a standardized rehabilitation therapy
* Written informed consent signed by the subject or next kin

Exclusion Criteria:

* Age < 18 years
* Pregnant and breastfeeding women
* Severe concomitant neurological (brain tumor, encephalitis, Parkinson disease, epilepsy prior to stroke onset) or mental disorders (psychiatric conditions such as schizophrenia, uncontrolled depression or bipolar disorder before stroke onset)
* Severe aphasia (i.e. unable to follow two-stage-commands)
* Pre-existing hemiparesis
* Documented history of dementia before index stroke
* Primary intracranial hematoma or subarachnoid hemorrhage
* Active implantable medical device (e.g., pacemaker, deep brain stimulator, cochlear implants, cerebral shunts)
* Metal cervical spine hardware or metallic implant near the stimulation site
* Modified Rankin scale (mRS) ≥ 2 prior to stroke onset
* Low heart rate (< 60 bpm)
* Severe vision and hearing problems
* Alcohol and drug abuse
* Active post-stroke delirium, unable to cooperate
* Type 1 and 2 diabetes mellitus
* Sore and diseased skin of the auricle
* Patients receiving any therapy (medication or otherwise) at study entry that would interfere with VNS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer-Motor-Assessment | Assessed <7 days and 6 weeks after admission at the Rheinburg Klinik.
  FMMA is a stroke-specific performance-based index of impairment. It has been designed to assess motor functioning, sensation, balance, joint range of motion and joint pain score in stroke survivors. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0 means "cannot perform"; 1 is "performs partially"; and 2 stands for "performs fully". In the present study, we will focus on the motor function score. It ranges from 0 (hemiplegia) to 100 points (normal motor function) and is divided into 66 points for the upper extremity and 34 points for the lower extremity. A difference of 5.25 points for the upper extremity and 6 points for the lower extremity are reported as minimal clinically important difference for the FMA.

SECONDARY OUTCOMES:
Consortium to Establish a Registry of Alzheimer's Disease (CERAD) | Assessed < 7 days and 6 weeks after admission to the Rheinburg Klinik.
  The CERAD neuropsychological test battery: includes 7 standardized subtests providing a comprehensive overview of a patient's cognitive performance. It is a proven tool in clinical practice and takes about 45 minutes to complete. The subtests are:
  * Semantic Fluency (Animals)
  * Boston Naming Test (BNT)
  * Learning and Memory Test
  * Constructional Praxis
  * Trail Making Tests (TMT) A and B
  * Phonemic Fluency (S-Words) The raw score is converted into standard scores (Z-scores), with Z-scores of -1 or lower considered indicative of cognitive impairment.
Montreal Cognitive Assessment (MoCA) | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The MoCA is a cognitive screening tool that requires the patient to complete 11 tasks assessing attention/concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The test takes approximately 10 minutes to administer with a maximum score of 30 points. Higher scores indicate better cognitive performance, a score of 26 or above is considered normal
Wechsler Adult Intelligence Scales (WAIS-IV) working memory subtests | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The WAIS-IV consists of different subtests and scales to measure intelligence in subjects aged 16 or older. The working memory subtests are used to assess short-term auditory memory and working memory. In the first test, participants are presented a sequence of numbers and asked to repeat them in the same order. In the "backward" condition, participants are asked to repeat the presented numbers in the reverse order. The first subtest measures short-term memory and attention, the second subtests is an indicator for working memory capacity and the ability to mentally manipulate information. The raw score is transformed into scaled scores, with values below 7 indicating a lower level of intelligence.
Digit Symbol Test | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The Digit Symbol Test is a well-established psychometric test paradigm which is used to measure general cognitive performance. Participants are asked to match numbers with corresponding symbols based on a key provided under time constraints. Number of correct matches are analyzed and are a measure of complex attention, working memory and associative learning. The Digit Symbol test is a widely used validated neuropsychological instrument that takes participants around 1-2 minutes to complete.
Stroop Color and Word Test | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The Stroop Test evaluates cognitive control and interference processing. Participants are asked to name the color of the ink used to print words, which can either match or conflict with the meaning of the word (for example the word "red" printed in blue color). The test measures executive functions, especially ability to inhibit cognitive interferences from the automatic process of reading. The Stroop Test takes around 5 minutes to complete.
Self-Report Measure for the Assessment of Emotion Regulation Skills (SEK-27) | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The SEK-27 is based on Berking's model of adaptive emotion regulation. Participants have to rate 27 items of 9 subscales (attention, clarity, bodily awareness, understanding, acceptance, resilience, self-support, willingness to confront, and regulation) on a 5-point Likert scale. The SEK-27 has a satisfactory internal consistency and test-retest reliability with a good reliability of the overall scale. The SEK-27 takes the participant around 3-10 minutes to complete. The score ranges from 27 to 135, with higher values indicating greater subjective emotional competence.
Emotion Regulation Questionnaire (ERQ) | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The Emotion Regulation Questionnaire (ERQ) assesses self-reported preferences for emotion regulation strategies. It consists of 10 items that are divided in two subscales (reappraisal and suppression). Higher scores indicate more frequent use of the respective strategy. Reappraisal is considered an adaptive strategy, while Suppression is regarded as a maladaptive strategy. There are no defined cutoff values, as the questionnaire is used to assess emotion regulation tendencies rather than classify them as dysfunctional.
Fatigue Scale for Motor and Cognitive Functions (FSMC) | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The FSMC, originally developed for multiple sclerosis, is a 20-item questionnaire assessing cognitive (e.g., "I have difficulty concentrating for extended periods") and physical fatigue (e.g., "I feel physically drained after minor physical exertion") on a five-point scale from "not at all" to "applies completely." The FSMC is also validated for assessing post-stroke fatigue. The score ranges from 20 to 100, with scores of 43 or higher Indicating fatigue-related impairment.
Pittsburgh Sleep Quality Index (PSQI) | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The PSQI is a questionnaire measuring sleep quality across several dimensions: subjective sleep quality, sleep latency, duration, efficiency, and disturbances. Responses are rated on a four-point scale, with a maximum score of 21 points. Higher scores indicate poorer sleep quality. The total score ranges from 0 to 21, with a score above 5 indicating impaired sleep quality.The PSQI is reliable and valid, taking about 5-10 minutes to complete.
Stroke-Specific Quality of Life Scale (SS-QOL) | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The SS-QOL evaluates health-related quality of life specifically designed for stroke survivors. This self-report questionnaire contains 49 items in 12 areas Energy, upper extremity function, Work/productivity, Mood, Self-care, Social roles, Family roles, Vision, Language, Thinking, Personality and functioning). Items are rated on a 5-point Likert scale. There are 3 different response sets i) "total help", score 1 to "no help needed", score 5; ii) "could not do it at all", score 1 to "no trouble at all", score 5; iii) "strongly agree", score 1 to "strongly disagree", score 5. Stroke survivors have to respond to each item using the corresponding response set. Scores of each item are added up to a total score ranging from 49 to 245. Higher scores indicate better functioning.
  Completion of the SS-QOL takes approximately 10-15 minutes.
Test of Attentional Performance (TAP) | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  Participants will complete the following sub-tests from the TAP:
  * TAP subtest Alertness: examines the participant's arousal level by measuring reaction times in tonic and phasic conditions. In the tonic condition, participants respond as quickly as possible to a cross appearing on the screen at random intervals (intrinsic alertness). In the phasic condition, the cross is preceded by a warning signal.
  * TAP subtest Go/NoGo: measures reaction inhibition. In this task, a cross or a plus appears on the screen and the participants are asked to respond only to the cross, suppressing the impulse to respond to the plus. This test assesses impulse control and inhibition ability.
  * TAP subtest Working Memory : measures the ability to control information flow and updating in working memory.
Action Research Arm Test (ARAT) | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The ARAT is a 19-item observational measure aimed at assessing the patients' ability to grasp (subscale with 6 items), grip (subscale with 4 items), pinch (subscale with 6 items) and perform gross movements (subscale with 3 items) with the upper extremity. The ARAT determines the patients' ability to handle objects that differ in size, weight and shape and thus, is an arm-specific measure of activity.
National Institutes of Health Stroke Scale (NIHSS) score | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The NIHSS score is a widely used and well validated score to objectively quantify the impairment and thus, to assess stroke severity in the acute phase of stroke and during follow-up. The NIHSS encompasses 11 items, each of which scores a particular ability between 0 (normal function) and 4 (seriously affected function). The scores from each item are added up to the total NIHSS score which ranges between 0 (no stroke symptoms) and a maximum score of 42 points (severe stroke). This score is done in a short time.
Modified Rankin Scale (mRS) | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of stroke survivors. The mRS is a 7-point scale ranging from 0 indicating no symptoms, 5 meaning severe disability and 6 standing for death.
Functional Independence Measure (FIM) | Assessed < 7 days and after 6 weeks after admission to the Rheinburg Klinik.
  The FIM is an assessment tool which allows to evaluate the functional status of patients throughout the rehabilitation process following stroke. The FIM score comprises a motor and cognitive domain. The motor domain consists of 13 items, the cognitive domain of 5 items. Each item is scored on a scale from 1 to 7, with 1 indicating complete dependence and 7 indicating complete independence in all areas. The total FIM score is calculated by adding the motor and cognitive scores, resulting in a total score between 18 and 126. A higher score indicates greater functional independence.
  It enables medical staff to track changes in the functional status of patients from the onset of rehabilitation care until discharge and follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Rheinburg Klinik, Walzenenhausen, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, ICF